CLINICAL TRIAL: NCT00527735
Title: A Randomized, Double Blind, Parallel, Three Arm Trial Evaluating the Efficacy and Safety of Ipilimumab (BMS-734016) in Combination With Paclitaxel/Carboplatin Compared to Paclitaxel/Carboplatin Alone in Previously Untreated Subjects With Lung Cancer
Brief Title: Phase II Study for Previously Untreated Subjects With Non Small Cell Lung Cancer (NSCLC) or Small Cell Lung Cancer (SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA184-041
Record Dates: First submitted 2007-09-07; First posted 2007-09-11 (Estimated); Results first posted 2012-07-16 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer; Small Cell Lung Cancer; Carcinoma, Non-Small-Cell Lung
Keywords: Non Small Cell Lung Cancer (NSCLC); Small Cell Lung Cancer (SCLC)
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Ipilimumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ipilimumab/ placebo + paclitaxel + carboplatin (concurrent) (Experimental)
  Interventions: Drug: Ipilimumab; Drug: Placebo; Drug: Paclitaxel; Drug: Carboplatin
- Ipilimumab/ placebo + paclitaxel + carboplatin (sequential) (Experimental)
  Interventions: Drug: Ipilimumab; Drug: Placebo; Drug: Paclitaxel; Drug: Carboplatin
- Ipilimumab placebo + paclitaxel + carboplatin (Active Comparator)
  Interventions: Drug: Placebo; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Ipilimumab — Ipilimumab, 10 mg/kg, administered as a single-dose, intravenously (IV), over 90 minutes depending on randomization every 3 weeks (up to 6 doses). Participants could receive additional maintenance ipilimumab at a dose of 10 mg/kg every 12 weeks starting 24 weeks after the first ipilimumab dose.
  Arms: Ipilimumab/ placebo + paclitaxel + carboplatin (concurrent); Ipilimumab/ placebo + paclitaxel + carboplatin (sequential)
Drug: Placebo — Matched placebo for ipilimumab administered as a single dose IV over 90 minutes every 3 weeks (up to 6 doses) as part of induction. Participants could also receive additional maintenance placebo administered IV over 90 minutes every 12 weeks starting 24 weeks after the first placebo dose.
Drug: Paclitaxel — 175 mg/m^2, administered as a single IV dose over 3 hours every 3 weeks (up to 6 doses). Dose modifications (reductions as well as delays) done as per product label.
Drug: Carboplatin — Area under the concentration curve (AUC)=6, administered as a single IV dose over 30 minutes every 3 weeks (up to 6 doses) as per randomization. Dose modifications (reductions as well as delays) done as per product label.

SUMMARY:
The purpose of the study is to determine whether ipilimumab given with paclitaxel/carboplatin has clinical benefit when compared with paclitaxel/carboplatin alone in patients with previously untreated lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed lung cancer (Stage IIIb/IV nonsmall-cell lung cancer or extensive stage small-cell lung cancer [SCLC])
* Measurable tumor lesion (as long as it is not located in a previously irradiated area) as defined by modified World Health Organization criteria
* Eastern Cooperative Oncology Group performance status of ≤1 at study entry
* Accessible for treatment and follow-up

Exclusion Criteria:

* Brain metastases
* Malignant pleural effusion
* Autoimmune disease
* Motor neuropathy of autoimmune origin
* SCLC-related paraneoplastic syndromes
* Any concurrent malignancy other than nonmelanoma skin cancer; carcinoma in situ of the cervix or breast; or prostate cancer treated with systemic therapy (participants with a previous malignancy but without evidence of disease for 5 years were allowed to enter the study)
* Prior systemic therapy for lung cancer. Prior radiation therapy or locoregional surgeries performed later than at least 3 weeks prior to randomization date were allowed.

  * Grade 2 peripheral neuropathy (motor or sensory)
* Known HIV or hepatitis B or C infection
* Chronic use of immunosuppressants and/or systemic corticosteroids (used in the management of cancer or noncancer-related illnesses). However, use of corticosteroids was allowed if used as premedication for paclitaxel infusion or for treating immune-related adverse events or adrenal insufficiencies.
* Inadequate hematologic function defined by an absolute neutrophil count <1,500/mm^3, a platelet count <100,000/mm^3, or hemoglobin level <9 g/dL.
* Inadequate hepatic function defined by a total bilirubin level >2.0 times the upper limit of normal (ULN), or ≥2.5 times the ULN if liver metastases are present, aspartate aminotransferase and alanine aminotransferase levels ≥2.5 times the ULN or ≥5 times the ULN if liver metastases are present.
* Inadequate renal function defined by a serum creatinine level ≥2.5 times the ULN
* Inadequate creatinine clearance defined as less than 50 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (66):
- United States (27):
  - Birmingham Hematology & Oncology Assoc. Llc, Birmingham, Alabama
  - Mayo Clinic, Scottsdale, Arizona
  - Acrc/Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Compassionate Cancer Care Medical Group, Corona, California
  - Compassionate Cancer Care Medical Group, Inc., Fountain Valley, California
  - The Angeles Clinic & Research Institute, Inc, Los Angeles, California
  - Oncology Care Medical Associates, Montebello, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - Sharp Clinical Oncology Research, San Diego, California
  - M D Anderson Cancer Center- Orlando, Orlando, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - University Of Chicago Medical Center, Chicago, Illinois
  - Local Institution, Park Ridge, Illinois
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - The John R. Marsh Cancer Center, Hagerstown, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - The Cancer Center, Minneapolis, Minnesota
  - Nevada Cancer Institute, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Local Institution, New York, New York
  - Cmc-Northeast/ Northeast Oncology Associates, Concord, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Hematology Oncology Consultants, Inc, Columbus, Ohio
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Guthrie Clinical Research, Sayre, Pennsylvania
  - Santee Hematology/Oncology, Sumter, South Carolina
  - Southwest Cancer Treatment And Research Center, Lubbock, Texas
- France (4):
  - Local Institution, Belfort
  - Local Institution, Caen
  - Local Institution, Marseille
  - Local Institution, Rennes
- Germany (10):
  - Local Institution, Bochum
  - Local Institution, Cologne
  - Local Institution, Coswig
  - Local Institution, Ebensfeld
  - Local Institution, Großhansdorf
  - Local Institution, Halle
  - Local Institution, Hamburg
  - Local Institution, Leipzig
  - Local Institution, Mainz
  - Local Institution, München
- India (5):
  - Local Institution, Hyderabad, Andhra Pradesh
  - Local Institution, Navrangpura, Ahmedabad, Gujarat
  - Local Institution, Manipal, Karnataka
  - Local Institution, Trivandrum, Kerala
  - Local Institution, Vellore
- Italy (3):
  - Local Institution, Genova
  - Local Institution, Siena
  - Local Institution, Torino
- Poland (4):
  - Local Institution, Gdansk
  - Local Institution, Krakow
  - Local Institution, Olsztyn
  - Local Institution, Szczecin
- Russia (7):
  - Local Institution, Arkhangelsk
  - Local Institution, Chelyabinsk
  - Local Institution, Ivanovo
  - Local Institution, Moscow
  - Local Institution, Pyatigorsk
  - Local Institution, Saint Petersburg
  - Local Institution, Sochi
- Ukraine (6):
  - Local Institution, Dnipropetrovsk
  - Local Institution, Donetsk
  - Local Institution, Kharkiv
  - Local Institution, Lviv
  - Local Institution, Ternopil
  - Local Institution, Uzhhorod

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 334 participants enrolled in this study, 331 received treatment. One patient with nonsmall-cell lung cancer, randomized to the sequential arm but mistakenly treated with concurrent therapy, is included in the sequential arm for efficacy results and in the concurrent arm for safety results.
Groups:
- Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 4 doses consisted of active ipilimumab with paclitaxel/carboplatin, and the last 2 doses consisted of placebo ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered intravenously (IV) as a single dose over 90 minutes. Participants who did not progress and did not experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until progressive disease (PD), drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Ipilimumab + Paclitaxel/Carboplatin (Sequential): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress and did not experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until PD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Placebo + Paclitaxel/Carboplatin: During induction, participants received up to 6 doses of placebo ipilimumab with paclitaxel/carboplatin every 3 weeks. Matched placebo for ipilimumab was administered as a single dose IV over 90 minutes every 3 weeks (up to 6 doses) as part of induction. Participants who did not progress or experience intolerable toxicity during the treatment phase could continue in the maintenance phase, receiving maintenance placebo administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose.
Period: Overall Study
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Started | 113 (Treated) | 109 (Treated) | 109 (Treated)
Completed | 5 (Still on treatment) | 2 (Still on treatment) | 2 (Still on treatment)
Not Completed | 108 | 107 | 107
Not completed — Disease progression | 47 | 61 | 53
Not completed — Death | 23 | 13 | 15
Not completed — Completed treatment in treatment phase | 14 | 13 | 18
Not completed — Adverse Event | 10 | 6 | 7
Not completed — Not identified | 5 | 5 | 5
Not completed — Withdrawal by Subject | 5 | 4 | 3
Not completed — No longer met study criteria | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 3
Not completed — Poor compliance or noncompliance | 0 | 1 | 1
Not completed — Completed treatment during maintenance | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin (concurrent). The initial 4 doses consisted of active ipilimumab with paclitaxel/carboplatin, and the last 2 doses consisted of placebo ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered intravenously (IV) as a single dose over 90 minutes every 3 weeks. Participants who experienced clinical benefit on treatment phase without intolerable toxicity were allowed to continue in the maintenance phase, receiving additional ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until immune-related progressive disease (irPD), drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin (sequential). The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes every 3 weeks. Participants who experienced clinical benefit on treatment phase without intolerable toxicity were allowed to continue in the maintenance phase, receiving additional ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until irPD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Placebo + Paclitaxel/Carboplatin: During induction, participants received up to 6 doses of placebo ipilimumab with paclitaxel/carboplatin. Matched placebo for ipilimumab was administered as a single dose IV over 90 minutes every 3 weeks (up to 6 doses) as part of induction. Participants who experienced clinical benefit on treatment phase without intolerable toxicity could continue in the maintenance phase, receiving maintenance placebo administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin | Total
Number analyzed (Participants) | 113 | 110 | 111 | 334
Age, Customized [Number; unit: Participants] — Age of participants who received treatment.
  Participants
    Younger than 65 years | 79 | 73 | 76 | 228
    65 years and older | 34 | 37 | 35 | 106
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 29 | 85
  Male | 86 | 81 | 82 | 249
Age Customized, by Disease Type [Number; unit: Participants] — NSCLC=nonsmall-cell lung cancer; SCLC=small-cell lung cancer
  Participants
    Younger than 65 years (NSCLC patients) | 44 | 44 | 40 | 128
    65 years and older (NSCLC patients) | 26 | 24 | 26 | 76
    Younger than 65 years (SCLC patients) | 35 | 29 | 36 | 100
    65 years and older (SCLC patients) | 8 | 13 | 9 | 30
Gender, by Disease Type [Number; unit: Participants] — NSCLC=nonsmall-cell lung cancer; SCLC=small-cell lung cancer
  Participants
    Female (NSCLC patients) | 17 | 19 | 17 | 53
    Male (NSCLC patients) | 53 | 49 | 49 | 151
    Female (SCLC patients) | 10 | 10 | 12 | 32
    Male (SCLC patients) | 33 | 32 | 33 | 98
Disease Stage at Study Entry [Number; unit: Participants] — NSCLC=nonsmall-cell lung cancer; SCLC=small-cell lung cancer. Staging of NSCLC is based on the findings of several clinical tests, including magnetic resonance imaging scans and fine needle biopsy. Stages range from 1 (best prognosis) to IV (worst prognosis). Stage I cancer is confined to the lung. Stages II and III cancers are locally advanced. Stage IV cancer has spread outside the lung to other organs. SCLC is staged using a 2-tiered system: Limited stage SCLC is confined to its area of origin in the lung and lumph nodes. Extensive-stage SCLC has spread beyond the lung to other organs.
  Participants
    Stage IIIB (NSCLC patients) | 11 | 7 | 17 | 35
    Stage IV (NSCLC patients) | 59 | 61 | 49 | 169
    Extensive (SCLC patients) | 43 | 42 | 44 | 129
    Recurrent disease (SCLC patients) | 0 | 0 | 1 | 1
Cell Type [Number; unit: Participants] — NSCLC=nonsmall-cell lung cancer; SCLC=small-cell lung cancer
  Participants
    Adenocarcinoma (NSCLC patients) | 35 | 30 | 38 | 103
    Bronchoalveolar carcinoma (NSCLC patients) | 1 | 1 | 0 | 2
    Large-cell carcinoma (NSCLC patients) | 6 | 11 | 7 | 24
    Other (NSCLC patients) | 6 | 4 | 3 | 13
    Squamous-cell carcinoma (NSCLC patients) | 21 | 21 | 15 | 57
    Unknown (NSCLC patients) | 1 | 1 | 3 | 5
    Other (SCLC patients) | 2 | 2 | 0 | 4
    Small-cell carcinoma (SCLC patients) | 41 | 38 | 45 | 124
    Unknown (SCLC patients) | 0 | 1 | 0 | 1
    Not reported (SCLC patients) | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Immune-related Progression-free Survival (irPFS) in Participants With Nonsmall-cell Lung Cancer (NSCLC) Per Immune-related Response Criteria (irRC)
Description: irPFS is defined as the time between the randomization date and date of immune-related Progressive Disease (irPD) (at least 25% increase percentage change in total tumor burden, including new lesions) or death, whichever occurs first. For patients with no recorded postbaseline tumor assessments, irPFS is censored at randomization. Participant who die without reported irPD are considered to have progressed on the date of death. For those who remain alive and have no irPD, irPFS is censored on the date of last evaluable tumor assessment. Independent review committee performed tumor assessment.
Time Frame: Tumor assessed at screening, every 6 weeks on treatment to Week 24, and every 12 weeks on maintenance until immune-related Progressive Disease (irPD) or death (of censored, maximum reached: 16.5 months)
Population: All participants with NSCLC who were randomized to a treatment group.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 4 doses consisted of active ipilimumab with paclitaxel/carboplatin, and the last 2 doses consisted of placebo ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered intravenously (IV) as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until immune-related progressive disease (irPD), drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Ipilimumab + Paclitaxel/Carboplatin (Sequential): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until irPD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 70 | 68 | 66
Months | 5.52 [4.17 to 6.74] | 5.68 [4.76 to 7.79] | 4.63 [4.14 to 5.52]
Statistical Analysis 1: Comparison: Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.1302, 1-sided log rank; Hazard Ratio (HR) = 0.806, 95% CI 2-sided [0.553 to 1.174]
Statistical Analysis 2: Comparison: Ipilimumab + Paclitaxel/Carboplatin (Sequential) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.0473, 1-sided log rank; Hazard Ratio (HR) = 0.724, 95% CI 2-sided [0.495 to 1.059]

2. Secondary Outcome: Progression-free Survival (PFS) in Participants With NSCLC Per Modified World Health Organization (mWHO) Criteria
Description: By mWHO criteria, PFS is defined as the time between the randomization date and the date of progression or death, whichever occurs first. For participants with no recorded postbaseline tumor assessment, PFS was censored at the day of randomization. A participant who died without reported prior progression was considered to have progressed on the date of death. For those who remain alive and have not progressed, PFS was censored on the date of last evaluable tumor assessment. Independent review committee performed tumor assessment.
Time Frame: Randomization date to date of progression or death (of censored, maximum reached: 13.6 months)
Population: All NSCLC participants who were randomized to a treatment group.
Measure: Mean (95% Confidence Interval); unit: Months
Groups:
- Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 4 doses consisted of active ipilimumab with paclitaxel/carboplatin, and the last 2 doses consisted of placebo ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress and did not experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until irPD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress and did not experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until PD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 70 | 68 | 66
Months | 4.11 [2.76 to 5.32] | 5.13 [4.17 to 5.72] | 4.21 [2.76 to 5.32]
Statistical Analysis 1: Comparison: Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.2502, One-sided log rank; Hazard Ratio (HR) = 0.882, 95% CI 2-sided [0.612 to 1.271]
Statistical Analysis 2: Comparison: Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.0240, One-sided log rank; Hazard Ratio (HR) = 0.691, 95% CI 2-sided [0.478 to 0.999]

3. Secondary Outcome: Overall Survival in Participants With NSCLC
Description: Overall Survival is defined as the time from the date of randomization until the date of death. For participants who have not died, Overall Survival was censored at the recorded last date of contact; participants with a missing recorded last date of contact were censored at the last date the participant was known to be alive.
Time Frame: Randomization date to date of death (of censored, maximum reached: 26.5 months)
Population: All NSCLC participants who were randomized to a treatment group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 70 | 68 | 66
Months | 9.69 [7.59 to 12.48] | 12.22 [9.26 to 14.39] | 8.28 [6.80 to 12.39]
Statistical Analysis 1: Comparison: Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.4759, 1-sided log rank; Hazard Ratio (HR) = 0.988, 95% CI 2-sided [0.669 to 1.460]
Statistical Analysis 2: Comparison: Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.2340, 1-sided log rank; Hazard Ratio (HR) = 0.866, 95% CI 2-sided [0.587 to 1.278]

4. Secondary Outcome: Best Overall Response Rate (BORR) Per mWHO Criteria in Participants With NSCLC and SCLC
Description: mWHO criteria define BORR as the number of patients with best overall response of Complete Response (CR) or Partial Response (PR), divided by the total number of participants in the data set (multiplied by 100 for percentage). CR=Complete disappearance of all index lesions; PR=decrease from baseline of >=50% in the sum of products of the 2 largest perpendicular diameters of all index lesions. Independent review committee performed tumor assessment.
Time Frame: Tumor assessment at screening, every 6 weeks on treatment to Week 24, and every 12 weeks on maintenance
Population: All participants who were randomized to a treatment group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 113 | 110 | 111
Percentage of participants
  BORR (mWHO criteria) NSCLC cohort (n=70, 68, 66) | 21.4 [12.5 to 32.29] | 32.4 [21.5 to 44.8] | 13.6 [6.4 to 24.3]
  BORR (mWHO criteria) SCLC cohort (n=43, 42, 45) | 32.6 [19.1 to 48.5] | 57.1 [41.0 to 72.3] | 48.9 [33.7 to 64.2]

5. Secondary Outcome: Immune-related Best Overall Response Rate (irBORR) Per irRC in Participants With NSCLC and Small-cell Lung Cancer (SCLC)
Description: irBORR=number of participants with irBORR of immune-related Complete Response (irCR) or immune-related Partial Response (irPR), divided by total participants in the data set. irCR=Complete disappearance of all index lesions. irPR=Decrease, relative to baseline, of 50% or greater in the sum of the products of the 2 largest perpendicular diameters of all index and of all new measurable lesions. Independent review committee performed the tumor assessments.
Time Frame: Tumor assessment at screening, every 6 weeks on treatment to Week 24, and every 12 weeks on maintenance
Population: All participants who were randomized to a treatment group.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 113 | 110 | 111
Percentage of participants
  irBORR ( irRC) NSCLC cohort (n=70, 68, 66) | 21.4 [12.5 to 32.29] | 32.4 [21.5 to 44.8] | 18.2 [9.8 to 29.6]
  irBORR (irRC) SCLC cohort (n=43, 42, 45) | 48.8 [33.3 to 64.5] | 71.4 [55.4 to 84.3] | 53.3 [37.9 to 68.3]

6. Secondary Outcome: Immune-related Disease Control Rate (irDCR) Per irRC and Disease Control Rate (DCR) Per mWHO Criteria in Participants With NSCLC and SCLC
Description: irDCR is defined as the proportion of participants whose immune-related best overall response is irPR, irCR, or immune-related Stable Disease (irSD) in the analysis data set. irSD=Does not meet criteria for irCR or irPR, in the absence of progressive disease. By mWHO criteria, DCR is defined as the proportion of participants whose best overall response is PR, CR, or SD in the analysis data set. SD=A decrease or tumor stabilization of 1 or more nonindex lesions. Independent review committee assessed response.
Time Frame: Tumor assessment at screening, every 6 weeks on treatment to Week 24, and every 12 weeks on maintenance until irPD, progressive disease, or death (maximum reached: 22 months)
Population: All participants who were randomized to a treatment group.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 113 | 110 | 111
Percent of participants
  irDCR (irRC) NSCLC cohort (n=70, 68, 66) | 70.0 [57.9 to 80.4] | 86.8 [76.4 to 93.8] | 81.8 [70.4 to 90.2]
  DCR (mWHO criteria) NSCLC cohort (n=70, 68, 66) | 57.1 [44.7 to 68.9] | 77.9 [66.2 to 87.1] | 72.7 [60.4 to 83.0]
  rDCR (irRC) SCLC cohort (n=43, 42, 45) | 81.4 [66.6 to 91.6] | 92.9 [80.5 to 98.5] | 95.6 [84.9 to 99.5]
  DCR (mWHO criteria) SCLC cohort (n=43, 42, 45) | 69.8 [53.9 to 82.8] | 81.0 [65.9 to 91.4] | 93.3 [81.7 to 98.6]

7. Secondary Outcome: Immune-related Duration of Response (irDoR) Per irRC and DoR Per mWHO Criteria in Participants With NSCLC and SCLC
Description: irDoR is defined as the time between the date of response of confirmed irCR or irPR and the date of irPD or death, whichever occurs first. For those participants who remain alive and did progress following response, irDoR was censored on the date of last evaluable tumor assessment. By mWHO criteria, DoR is defined as the time between the date of response of confirmed CR or PR and the date of PD or death, whichever occurs first. For those who remain alive and did not progress following response, DoR was censored on the date of last evaluable tumor assessment.
Time Frame: Date of irCR or irPR to date of irPD or death (maximum reached: 14.2 months)
Population: All participants who were randomized to a treatment group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 113 | 110 | 111
Months
  irDoR (irRC) NSCLC cohort (n=70, 63, 62) | 6.70 [4.21 to 8.51] | 5.55 [4.27 to 6.74] | 4.01 [4.01 to 5.72]
  DoR (mWHO criteria) NSCLC cohort (n=70, 63, 62) | 5.42 [4.21 to 7.43] | 5.55 [4.27 to 6.74] | 4.01 [3.94 to 5.59]
  irDoR (irRC) SCLC cohort (n=43, 42, 45) | 5.95 [4.53 to 10.8] | 5.78 [4.44 to 6.67] | 4.21 [3.91 to 6.41]
  DoR (mWHO criteria) SCLC cohort (n=43, 42, 45) | 7.62 [4.90 to 11.1] | 5.78 [3.94 to 6.57] | 4.21 [3.91 to 5.95]

8. Secondary Outcome: Number of Participants With NSCLC Who Have Death as Outcome, Serious Adverse Events (SAEs), Drug-related SAEs, Adverse Events (AEs), AEs Leading to Discontinuation, and Drug-related AEs by Worst Common Terminology Criteria (CTC) Grade
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Drug-related=possibly, probably, or certainly related to and of unknown relationship to study drug. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Life-threatening or disabling, Gr 5=Death.
Time Frame: Weeks 4, 7, 10, 16, 19, and 24; at end of treatment; and at follow-up (70 days from last dose)
Population: All participants with NSCLC who received at least 1 dose of blinded active or placebo ipilimumab with or without paclitaxel/carboplatin. One NSCLC participant randomized to the sequential arm is included in the concurrent arm for safety evaulations.
Measure: Number; unit: Participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 71 | 67 | 65
Participants
  Deaths (total) | 52 | 50 | 51
  Deaths within 30 days of last dose of study drug | 11 | 7 | 8
  Deaths within 70 days of last dose of study drug | 21 | 16 | 18
  SAEs (total) | 49 | 36 | 33
  SAEs, Grade 3 | 17 | 16 | 9
  SAEs, Grade 4 | 10 | 4 | 5
  SAEs, Grade 5 | 20 | 15 | 18
  SAEs, Drug-related | 20 | 13 | 11
  SAEs, Drug-related Grade 5 | 2 | 1 | 2
  AEs leading to discontinuation (disc) (total) | 28 | 19 | 15
  AEs leading to disc, Drug-related (all) | 16 | 7 | 8
  AEs leading to disc, Drug-related Grade 3 | 9 | 6 | 4
  AEs leading to disc, Drug-related Grade 4 | 1 | 0 | 0
  AEs leading to disc, Drug-related Grade 5 | 1 | 0 | 1
  AEs (total) | 71 | 64 | 64
  AEs, Grades 3 and 4 | 40 | 36 | 26
  AEs, Drug-related Any Grade | 56 | 56 | 54
  AEs, Drug-related Grades 3 and 4 | 29 | 26 | 24
  AEs, Drug-related Grade 5 | 2 | 1 | 2

9. Secondary Outcome: Percentage of Participants With NSCLC Who Have Abnormalities in On-study Hematology Laboratory Test Results by Worst CTC Grade
Description: CTC, Version 3 used to assess parameters. LLN=lower limit of normal. CTC criteria: ANC=absolute neutrophil count. White blood cells Grade (Gr) 1:<LLN to 3.0*10^9/L, Gr 2:<3.0 to 2.0*10^9/L, Gr 3:<2.0 to 1.0*10^9/L, Gr 4:<1.0*10^9/L. ANC Gr 1:<LLN to 1.5*10^9/L, Gr 2:<1.5 to 1.0*10^9/L, Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L. Platelet count Gr 1:LLN to 75.0*10^9/L, Gr 2:<75.0 to 50.0*10^9/L, Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0 to 10^9/L. Hemoglobin Gr 1:<LLN to 10.0 g/dL, Gr 2:<10.0 to 8.0 g/dL, Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL.
Time Frame: At screening; predose Day 1; and Weeks 4, 7, 10, 13, 16, 19, and 24; and every 12 weeks on maintenance until disease progression, study closure, or withdrawal of consent
Population: All participants with NSCLC who received at least 1 dose of ipilimumab/placebo and/or chemotherapy and had at least 1 on-study hematology test result available. One NSCLC participant randomized to the sequential arm is included in the concurrent arm for safety evaulations.
Measure: Number; unit: Percentage of participants
Groups:
- Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 4 doses consisted of active ipilimumab with paclitaxel/carboplatin, and the last 2 doses consisted of placebo ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until irPD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until irPD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 71 | 67 | 65
Percentage of participants
  White blood cell count, Grades 3 and 4 | 7.7 | 6.2 | 3.2
  Hemoglobin, Any grade | 90.8 | 98.5 | 90.2
  Hemoglobin, Grades 3 and 4 | 10.8 | 6.2 | 6.3
  ANC, Grades 3 and 4 | 7.7 | 1.5 | 9.5
  Platelets, Grades 3 and 4 | 1.5 | 3.1 | 9.5

10. Secondary Outcome: irPFS in Participants With SCLC Per irRC
Description: IRC performed TA.
Time Frame: Randomization date to date of irPD or death (maximum reached: 22 months)
Population: All participants with SCLC who were randomized to a treatment group.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 43 | 42 | 45
Months | 5.68 [5.19 to 6.87] | 6.44 [5.29 to 7.75] | 5.26 [4.67 to 5.72]
Statistical Analysis 1: Comparison: Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.1098, 1-sided log rank; Hazard Ratio (HR) = 0.751, 95% CI 2-sided [0.475 to 1.188]
Statistical Analysis 2: Comparison: Ipilimumab + Paclitaxel/Carboplatin (Sequential) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.0282, 1-sided log rank; Hazard Ratio (HR) = 0.640, 95% CI 2-sided [0.403 to 1.1016]

11. Secondary Outcome: Number of Participants With NSCLC Who Have Abnormalities in On-Study Liver Function Test Results By Worst CTC Grade
Description: ULN=Upper limit of normal among all laboratory ranges. ALT=alanine transaminase; AST=aspartate aminotransferase; ALK=alkaline phosphatase. CTC grade criteria: ALT Grade 1:>ULN to 2.5*ULN; Grade 2: >2.5 to 5.0*ULN; Grade 3: >5.0 to 20.0*ULN; Grade 4: >20.0*ULN. AST Grade 1: >ULN to 2.5*ULN; Grade 2: >2.5 to 5.0*ULN; Grade 3: >5.0 to 20.0*ULN; Grade 4: >20.0*ULN. Total bilirubin Grade 1: >ULN to 1.5*ULN; Grade 2: >1.5 to 3.0*ULN; Grade 3: >3.0 to 10.0*ULN; Grade 4: >10.0*ULN. ALK (U/L) G1:>ULN to 2.5*ULN, G2:>2.5 to 5.0*ULN, G3:>5.0 to 20.0*ULN, G4:>20.0*ULN.
Time Frame: At screening; predose Day 1; Weeks 4, 7, 10, 13, 16, 19, and 24; and every 12 weeks on maintenance until disease progression, study closure, or withdrawal of consent
Population: All participants with NSCLC who received at least 1 dose of ipilimumab and/or chemotherapy and had at least 1 on-study liver function measurement available. One NSCLC participant randomized to the sequential arm is included in the concurrent arm for safety evaulations.
Measure: Number; unit: Participants
Groups:
- Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until PD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 65 | 65 | 62
Participants
  Alanine aminotransferase (ALT), Grade 1 | 24 | 15 | 19
  ALT, Grade 2 | 2 | 4 | 3
  ALT, Grades 3 and 4 | 1 | 1 | 1
  Aspartate aminotransferase (AST), Grade 1 | 16 | 18 | 20
  AST, Grade 2 | 0 | 2 | 0
  AST, Grades 3 and 4 | 1 | 1 | 1
  Total bilirubin, Grade 1 | 1 | 3 | 2
  Total bilirubin, Grade 2 | 3 | 2 | 1
  Total bilirubin, Grades 3 and 4 | 0 | 0 | 0
  Alkaline phosphatase, Grade 1 | 24 | 28 | 24
  Alkaline phosphatase, Grade 2 | 1 | 2 | 3
  Alkaline phosphatase, Grades 3 and 4 | 0 | 1 | 1

12. Secondary Outcome: Number of Participants With NSCLC Who Had Abnormalities in Vital Sign Measurements and Physical Examination Findings
Description: Vital signs measurements consisted of systolic and diastolic blood pressure, heart rate, temperature, and respiratory rate. Physical examinations assessed weight, height, performance status, and body surface area.
Time Frame: At screening; Day 1; Weeks 4, 7, 10, 13, 16, and 24; and every 12 weeks on maintenance until disease progression, study closure, or withdrawal of consent
Population: All participants with NSCLC who received at least 1 dose of ipilimumab/placebo and/or chemotherapy and had at least 1 on-study measurement available.One NSCLC participant randomized to the sequential arm is included in the concurrent arm for safety evaulations.
Measure: Number; unit: Participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 71 | 67 | 65
Participants
  Vital sign measurements | 0 | 0 | 0
  Physical examination findings | 0 | 0 | 0

13. Secondary Outcome: Percentage of Participants With NSCLC Who Have Abnormalities in Pancreatic Enzyme Clinical Laboratory Test Results by Worst CTC Grade
Description: ULN=upper limit of normal. Lipase (U/L) Gr 1: 1.1 to 1.39*ULN; Gr 2: >1.5 to 2.0*ULN; Gr 3: 2.5 to 5; Gr 4: 5*ULN. Amylase (U/L) Gr 1: >ULN to 1.5*ULN; Grade 2 >1.5 to 2.0*ULN, Grade 3 >2.0 to 5.0*ULN, Grade 4 >5.0*ULN. Creatine (mg/dL) Grade 1: >ULN to 1.5*ULN, Gr 2: 1.5 to 3.0*ULN, Gr 3: >3.0 to 6.0*ULN, Gr 4: >6.0*ULN.
Time Frame: At screening; predose Day 1; Weeks 4, 7, 10, 13, 16, 19, and 24; and at end of treatment
Population: All participants with NSCLC who received at least 1 dose of ipilimumab/placebo and/or chemotherapy and had at least 1 on-study pancreatic enzyme laboratory test measurement available. One NSCLC participant randomized to the sequential arm is included in the concurrent arm for safety evaulations.
Measure: Number; unit: Percentage of participants
Groups:
- Ipilimumab + Paclitaxel/Carboplatin (Sequential): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until PD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 71 | 67 | 65
Percentage of participants
  Lipase, Grades 3 and 4 | 7.7 | 6.2 | 3.2
  Amylase, Grades 3 and 4 | 1.5 | 4.6 | 1.6

14. Secondary Outcome: Number of Participants With NSCLC Who Have Positive Human Antihuman Antibody (HAHA) Status Postbaseline
Description: An electrochemilumiluminescent immunoassay was used to detect HAHA antibodies to ipilimumab in human serum. Baseline, either negative or positive, is the maximum of all measurements closest and prior to the first ipilimumab dose. Positive status postbaseline=participants with an increase in HAHA measurement from baseline.
Time Frame: Day 1; Weeks 4, 7, 10, 13, 16, 19, and 24; and at end of treatment
Population: Participants with at least 1 HAHA measurement prior to and at least 1 after the first ipilimumab dose and with an increase in HAHA measurement from baseline.
Measure: Number; unit: Participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential)
Number analyzed (Participants) | 61 | 56
Participants | 2 | 1

15. Secondary Outcome: Number of Participants With SCLC With Death as Outcome, Serious Adverse Events (SAEs), Drug-related SAEs, Adverse Events (AEs), AEs Leading to Discontinuation, Drug-related AEs by Worst CTC Grade
Description: as for outcome 8
Time Frame: Weeks 4, 7, 10, 16, 19, and 24; at end of treatment; and at follow-up (70 days from last dose)
Population: All participants with SCLC who received at least 1 dose of blinded active or placebo ipilimumab with or without paclitaxel/carboplatin.
Measure: Number; unit: Participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 42 | 42 | 44
Participants
  Deaths (total) | 37 | 31 | 35
  Deaths within 30 days of last dose of study drug | 6 | 2 | 1
  Deaths within 70 days of last dose of study drug | 13 | 7 | 8
  SAEs (total) | 25 | 21 | 20
  SAEs, Grade 3 | 7 | 6 | 4
  SAEs, Grade 4 | 3 | 4 | 4
  SAEs, Grade 5 | 12 | 7 | 7
  SAEs, Drug-related | 10 | 12 | 6
  SAEs, Drug-related Grade 5 | 1 | 0 | 0
  AEs leading to discontinuation (disc) (total) | 14 | 13 | 12
  AEs leading to disc, Drug-related (all) | 9 | 7 | 7
  AEs leading to disc, Drug-related Grade 3 | 3 | 3 | 4
  AEs leading to disc, Drug-related Grade 4 | 2 | 2 | 0
  AEs leading to disc, Drug-related Grade 5 | 1 | 0 | 0
  AEs (total) | 41 | 40 | 43
  AEs, Grades 3 and 4 | 19 | 22 | 19
  AEs, Grade 5 | 12 | 7 | 7
  AEs, Drug-related (all) | 36 | 40 | 40
  AEs, Drug-related,Grades 3 and 4 | 18 | 21 | 13
  AEs, Drug-related, Grade 5 | 1 | 0 | 0

16. Secondary Outcome: Number of Participants With SCLC Who Have Abnormalities in On-study Hematology Laboratory Test Results by Worst CTC Grade
Description: CTC, Version 3 used to assess parameters. LLN=lower limit of normal. CTC criteria: ANC=absolute neutrophil count. White blood cells Gr 1:<LLN to 3.0*10^9/L, Gr 2:<3.0 to 2.0*10^9/L, Gr 3:<2.0 to 1.0*10^9/L, Gr 4:<1.0*10^9/L. ANC Gr 1:<LLN to 1.5*10^9/L, Gr 2:<1.5 to 1.0*10^9/L, Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L. Platelet count Gr 1:LLN to 75.0*10^9/L, Gr 2:<75.0 to 50.0*10^9/L, Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0 to 10^9/L. Hemoglobin Gr 1:<LLN to 10.0 g/dL, Gr 2:<10.0 to 8.0 g/dL, Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL.
Time Frame: At screening, predose Day 1, and Weeks 4, 7, 10, 13, 16, 19, 24, and at end of treatment
Population: All participants with SCLC who received at least 1 dose of ipilimumab and/or chemotherapy and had at least 1 on-study hematology test result available.
Measure: Number; unit: Participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 42 | 42 | 44
Participants
  White blood cells, Grade 1 (n=39, 42, 43) | 7 | 11 | 13
  White blood cells, Grade 2 (n= 39, 42, 43) | 10 | 9 | 7
  White blood cells, Grades 3 (n= 39, 42, 43) | 0 | 2 | 0
  White blood cells, Grade 4 (n= 39, 42, 43) | 0 | 0 | 0
  Absolute neutrophil count, Grade 1 (n= 39, 42, 43) | 8 | 8 | 8
  Absolute neutrophil count, Grade 2 (n= 39, 42, 43) | 8 | 9 | 91
  Absolute neutrophil count, Grade 3 (n= 39, 42, 43) | 2 | 2 | 1
  Absolute neutrophil count, Grade 4 (n= 39, 42, 43) | 1 | 2 | 0
  Platelet count, Grade 1 (n= 39, 42, 43) | 15 | 18 | 23
  Platelet count, Grade 2 (n= 39, 42, 43) | 2 | 3 | 3
  Platelet count, Grade 3 (n= 39, 42, 43) | 1 | 2 | 1
  Platelet count, Grade 4 (n= 39, 42, 43) | 0 | 1 | 0
  Hemoglobin, Grade 1 (n= 39, 42, 43) | 26 | 24 | 25
  Hemoglobin, Grade 2 (n= 39, 42, 43) | 8 | 10 | 11
  Hemoglobin, Grade 3 (n= 39, 42, 43) | 2 | 2 | 3
  Hemoglobin, Grade 4 (n= 39, 42, 43) | 0 | 2 | 0

17. Secondary Outcome: Number of Participants With SCLC Who Have Abnormalities in Liver Function Test Results by Worst CTC Grade
Description: ALT=alanine aminotransferase; AST=aspartate aminotransferase; ALK=alkaline phosphatase. ULN=Upper limit of normal among all laboratory ranges. CTC grade criteria: ALT Grade 1:>ULN to 2.5*ULN; Grade 2: >2.5 to 5.0*ULN; Grade 3: >5.0 to 20.0*ULN; Grade 4: >20.0*ULN. AST Grade 1: >ULN to 2.5*ULN; Grade 2: >2.5 to 5.0*ULN; Grade 3: >5.0 to 20.0*ULN; Grade 4: >20.0*ULN. Total bilirubin Grade 1: >ULN to 1.5*ULN; Grade 2: >1.5 to 3.0*ULN; Grade 3: >3.0 to 10.0*ULN; Grade 4: >10.0*ULN. ALK (U/L) G1:>ULN to 2.5*ULN, G2:>2.5 to 5.0*ULN, G3:>5.0 to 20.0*ULN, G4:>20.0*ULN.
Time Frame: At screening; predose Day 1; Weeks 4, 7, 10, 13, 16, 19, and 24; and at end of treatment
Population: All participants with SCLC who received at least 1 dose of ipilimumab/placebo and/or chemotherapy and had at least 1 on-study liver function test result available.
Measure: Number; unit: Participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 42 | 42 | 44
Participants
  ALT, Grade 1 | 12 | 12 | 8
  ALT, Grade 2 | 2 | 3 | 1
  ALT, Grades 3 & 4 | 7 | 2 | 0
  AST, Grade 1 | 11 | 13 | 12
  AST, Grade 2 | 4 | 1 | 2
  AST, Grades 3 & 4 | 5 | 3 | 0
  Total bilirubin, Grade 1 | 4 | 5 | 3
  Total bilirubin, Grade 2 | 1 | 0 | 0
  Total bilirubin, Grades 3 & 4 | 1 | 0 | 0
  ALK, Grade 1 | 15 | 14 | 16
  ALK, Grade 2 | 1 | 3 | 2
  ALK, Grades 3 & 4 | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants With SCLC Who Have Abnormalities in Pancreatic Enzyme and Other Clinical Laboratory Test Results by Worst CTC Grade
Description: ULN=upper limit of normal. Lipase (U/L) Grade (Gr) 1: 1.1 to 1.39*ULN; Gr 2: >1.5 to 2.0*ULN; Gr 3: 2.5 to 5; Gr 4: 5*ULN. Amylase (U/L) Gr 1: >ULN to 1.5*ULN; Gr 2 >1.5 to 2.0*ULN, Gr 3 >2.0 to 5.0*ULN, Gr 4 >5.0*ULN. Creatine (mg/dL) Gr 1: >ULN to 1.5*ULN, Gr 2: 1.5 to 3.0*ULN, Gr 3: >3.0 to 6.0*ULN, Gr 4: >6.0*ULN.
Time Frame: At screening, predose Day 1, and Weeks 4, 7, 10, 13, 16, 19, 24, and at end of treatment
Population: All participants with SCLC who received at least 1 dose of ipilimumab and/or chemotherapy and had at least 1 on-study pancreatic enzyme or other laboratory test measurement available.
Measure: Number; unit: Percentage of participants
Groups:
- Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin (concurrent). The initial 4 doses consisted of active ipilimumab with paclitaxel/carboplatin, and the last 2 doses consisted of placebo ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered intravenously (IV) as a single dose over 90 minutes every 3 weeks as part of induction. Participants could also receive additional maintenance ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose.
- Ipilimumab + Paclitaxel/Carboplatin (Sequential): During induction, participants received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin (sequential). The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes every 3 weeks as part of induction. Participants could also receive additional maintenance ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose.
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 42 | 42 | 44
Percentage of participants
  Lipase, Grades 3 and 4 | 7.7 | 16.7 | 11.6
  Amylase, Grades 3 and 4 | 5.1 | 4.8 | 4.7
  Creatinine, Grades 3 and 4 | 0 | 0 | 0

19. Secondary Outcome: Progression-free Survival (PFS) in Participants With SCLC Per mWHO Criteria
Description: By mWHO criteria, PFS is defined as the time between the randomization date and the date of progression or death, whichever occurs first. For participants with no recorded postbaseline tumor assessment, PFS was censored at the day of randomization. A participant who died without reported prior progression was considered to have progressed on the date of death. For those who remain alive and have not progressed, PFS was censored on the date of last evaluable tumor assessment.
Time Frame: Randomization date to date of progression or death (of censored, maximum reached: 22 months)
Population: All participants with SCLC who were randomized to a treatment group.
Measure: Mean (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 43 | 42 | 45
Months | 3.89 [2.89 to 5.85] | 5.22 [4.14 to 6.57] | 5.19 [4.40 to 5.59]
Statistical Analysis 1: Comparison: Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.3846, 1-sided Log Rank; Hazard Ratio (HR) = 0.933, 95% CI 2-sided [0.588 to 1.481]
Statistical Analysis 2: Comparison: Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.3700, 1-sided Log Rank; Hazard Ratio (HR) = 0.927, 95% CI 2-sided [0.591 to 1.453]

20. Secondary Outcome: Number of Participants With SCLC Who Had Abnormalities in Vital Sign Measurements and Physical Examination Findings
Description: as for outcome 12
Time Frame: Predose Day 1; Weeks 4, 7, 10, 13, 16, and 24; and every 12 weeks on maintenance until end of treatment
Population: All participants with SCLC who received at least 1 dose of ipilimumab/placebo and/or chemotherapy and had at least 1 on-study measurement available.
Measure: Number; unit: Participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 42 | 42 | 44
Participants
  Vital sign measurements | 0 | 0 | 0
  Physical examination findings | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With SCLC Who Have Positive HAHA Status Postbaseline
Description: as for outcome 14
Time Frame: Day 1; Weeks 4, 7, 10, 13, 16, 19, and 24; and at end of treatment
Population: Participants with SCLC who had at least 1 HAHA measurement prior to and at least 1 after the first ipilimumab dose and with an increase in HAHA measurement from baseline.
Measure: Number; unit: Participants
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Ipilimumab + Paclitaxel/Carboplatin (Sequential)
Number analyzed (Participants) | 38 | 41
Participants
  Positive at any timepoint (n=42, 42) | 2 | 3
  Positive postbaseline (n=38, 41) | 2 | 0

22. Secondary Outcome: Overall Survival in Participants With SCLC
Description: as for outcome 3
Time Frame: Randomization date to date of death (of censored, maximum reached: 22 months)
Population: All participants with SCLC who were randomized to a treatment group.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) | Placebo + Paclitaxel/Carboplatin
Number analyzed (Participants) | 43 | 42 | 45
Months | 3.89 [2.89 to 5.85] | 5.22 [4.14 to 6.57] | 5.19 [4.40 to 5.59]
Statistical Analysis 1: Comparison: Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.4132, 1-sided Log Rank; Hazard Ratio (HR) = 0.947, 95% CI 2-sided [0.585 to 1.536]
Statistical Analysis 2: Comparison: Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) vs Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) vs Placebo + Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.1287, 1-sided Log Rank; Hazard Ratio (HR) = 0.753, 95% CI 2-sided [0.461 to 1.232]

ADVERSE EVENTS:
Groups:
- Ipilimubab+Paclitaxel/Carboplatin (Concurrent) NSCLC: During induction, participants with nonsmall-cell lung cancer (NSCLC) received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 4 doses consisted of active ipilimumab with paclitaxel/carboplatin, and the last 2 doses consisted of placebo ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered intravenously (IV) as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered intravenously (IV) over 90 minutes every 12 weeks starting 24 weeks after the first dose until immune-related progressive disease (irPD), drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Placebo/Ipilimumab+ Paclitaxel/Carboplatin (Sequential) NSCLC: During induction, participants with NSCLC received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until irPD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Placebo + Paclitaxel/Carboplatin NSCLC: During induction, participants with NSCLC received up to 6 doses of placebo ipilimumab with paclitaxel/carboplatin every 3 weeks. Matched placebo for ipilimumab was administered as a single dose IV over 90 minutes every 3 weeks (up to 6 doses) as part of induction. Participants who did not progress or experience intolerable toxicity during the treatment phase could continue in the maintenance phase, receiving maintenance placebo administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose.
- Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) SCLC: During induction, participants with small-cell lung cancer (SCLC) received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 4 doses consisted of active ipilimumab with paclitaxel/carboplatin, and the last 2 doses consisted of placebo ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until irPD, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) SCLC: During induction, participants with SCLC received up to 6 doses of blinded ipilimumab with paclitaxel/carboplatin on a 3-week schedule. The initial 2 doses consisted placebo ipilimumab with paclitaxel/carboplatin followed by 4 doses of active ipilimumab with paclitaxel/carboplatin. Ipilimumab, 10 mg/kg, was administered IV as a single dose over 90 minutes. Participants who did not progress or experience intolerable toxicity during the treatment phase were allowed to continue in the maintenance phase, receiving additional (blinded) ipilimumab at a dose of 10 mg/kg administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose until progressive disease, drug intolerance, withdrawal of consent, pregnancy, death, loss to follow up, or study closure.
- Placebo + Paclitaxel/Carboplatin SCLC: During induction, participants with SCLC received up to 6 doses of placebo ipilimumab with paclitaxel/carboplatin every 3 weeks. Matched placebo for ipilimumab was administered as a single dose IV over 90 minutes every 3 weeks (up to 6 doses) as part of induction. Participants who did not progress or experience intolerable toxicity during the treatment phase could continue in the maintenance phase, receiving maintenance placebo administered IV over 90 minutes every 12 weeks starting 24 weeks after the first dose.
Arm/Group | Ipilimubab+Paclitaxel/Carboplatin (Concurrent) NSCLC | Placebo/Ipilimumab+ Paclitaxel/Carboplatin (Sequential) NSCLC | Placebo + Paclitaxel/Carboplatin NSCLC | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) SCLC | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) SCLC | Placebo + Paclitaxel/Carboplatin SCLC
Serious Adverse Events (participants affected / at risk) | 49/71 | 36/67 | 33/65 | 25/42 | 21/42 | 20/44
Other Adverse Events (participants affected / at risk) | 63/71 | 63/67 | 59/65 | 36/42 | 39/42 | 41/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimubab+Paclitaxel/Carboplatin (Concurrent) NSCLC (N=71) | Placebo/Ipilimumab+ Paclitaxel/Carboplatin (Sequential) NSCLC (N=67) | Placebo + Paclitaxel/Carboplatin NSCLC (N=65) | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) SCLC (N=42) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) SCLC (N=42) | Placebo + Paclitaxel/Carboplatin SCLC (N=44)
ANAEMIA (Blood and lymphatic system disorders) | 4 | 4 | 1 | 0 | 2 | 2
ARTERIAL THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
AUTOIMMUNE HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
GASTROENTERITIS SHIGELLA (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
HYPOPITUITARISM (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
MALIGNANT PLEURAL EFFUSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
METASTATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 0 | 1 | 1 | 1
SIALOADENITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 2 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 2 | 2 | 4 | 0 | 0 | 0
ERYSIPELAS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
ERYTHEMA MULTIFORME (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 | 1 | 2 | 1 | 0 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPOTENSION (Vascular disorders) | 1 | 1 | 2 | 1 | 0 | 1
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
BRONCHITIS CHRONIC (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
CACHEXIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
COLITIS (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
DYSARTHRIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 2 | 1 | 0 | 2 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
HYDROCEPHALUS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
HYPOPHYSITIS (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
MULTI-ORGAN FAILURE (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
PERICARDIAL EFFUSION MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
PYREXIA (General disorders) | 1 | 3 | 0 | 4 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
TACHYARRHYTHMIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
THROMBOPHLEBITIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 2
ASTHENIA (General disorders) | 1 | 1 | 1 | 1 | 0 | 0
ATAXIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
CELLULITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
EPILEPSY (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
FEBRILE INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
ILEAL PERFORATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
LUNG CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | 0
NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 3 | 4 | 2 | 3
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 0 | 3 | 0 | 3 | 3
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
TOXIC EPIDERMAL NECROLYSIS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0 | 2 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
CERVICAL CORD COMPRESSION (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
DERMATITIS EXFOLIATIVE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 1 | 1 | 1 | 0 | 0 | 0
MACULAR CYST (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
NON-SMALL CELL LUNG CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0 | 0
PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
SALIVARY GLAND CALCULUS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 2 | 0 | 3 | 1
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
VERTIGO (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
ANAPHYLACTIC REACTION (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
ANGINA PECTORIS (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
CONVULSION (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 7 | 5 | 4 | 1 | 2 | 1
DUODENAL ULCER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
ENTERITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
GASTROINTESTINAL PERFORATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
GRAND MAL CONVULSION (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
MEDIASTINAL DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
MENINGITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
OESOPHAGEAL DISORDER (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
PANCREATITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
PATHOLOGICAL FRACTURE (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
PERIPHERAL SENSORIMOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0
VENOUS THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
ABDOMINAL HERNIA (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
BASAL GANGLIA HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
BILIARY COLIC (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0
DEATH (General disorders) | 2 | 4 | 2 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 2 | 1 | 1
EROSIVE OESOPHAGITIS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
FATIGUE (General disorders) | 1 | 2 | 1 | 1 | 1 | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
HEPATOTOXICITY (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0
LOCALISED OEDEMA (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4 | 5 | 4 | 6 | 5
MONOPLEGIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
NEUROPATHY PERIPHERAL (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
SUDDEN DEATH (General disorders) | 0 | 2 | 0 | 0 | 0 | 0
TRACHEO-OESOPHAGEAL FISTULA (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
ACIDOSIS (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
DISEASE PROGRESSION (General disorders) | 5 | 1 | 4 | 1 | 0 | 1
DROWNING (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0
ICHTHYOSIS (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
LUNG DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
OCCIPITAL NEURALGIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
PLEURAL INFECTION BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 5 | 2 | 2 | 0 | 0 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimubab+Paclitaxel/Carboplatin (Concurrent) NSCLC (N=71) | Placebo/Ipilimumab+ Paclitaxel/Carboplatin (Sequential) NSCLC (N=67) | Placebo + Paclitaxel/Carboplatin NSCLC (N=65) | Ipilimumab/Placebo + Paclitaxil/Carboplatin (Concurrent) SCLC (N=42) | Placebo/Ipilimumab + Paclitaxel/Carboplatin (Sequential) SCLC (N=42) | Placebo + Paclitaxel/Carboplatin SCLC (N=44)
ANAEMIA (Blood and lymphatic system disorders) | 22 | 15 | 19 | 13 | 12 | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 18 | 11 | 10 | 13 | 23 | 15
DIZZINESS (Nervous system disorders) | 9 | 7 | 5 | 1 | 2 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 22 | 27 | 22 | 11 | 13 | 13
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 7 | 9 | 5 | 5 | 6 | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 3 | 2 | 1 | 1 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 6 | 2 | 4 | 4 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 13 | 10 | 11 | 9 | 8 | 11
DEHYDRATION (Metabolism and nutrition disorders) | 4 | 5 | 3 | 1 | 2 | 3
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 5 | 1 | 2 | 0
HYPOTENSION (Vascular disorders) | 4 | 1 | 8 | 0 | 2 | 0
WEIGHT DECREASED (Investigations) | 10 | 10 | 5 | 6 | 7 | 3
CONSTIPATION (Gastrointestinal disorders) | 13 | 10 | 15 | 5 | 4 | 9
DYSPHAGIA (Gastrointestinal disorders) | 1 | 5 | 3 | 1 | 1 | 2
ERYTHEMA (Skin and subcutaneous tissue disorders) | 4 | 2 | 1 | 0 | 0 | 0
HAEMOGLOBIN DECREASED (Investigations) | 3 | 5 | 2 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 8 | 9 | 8 | 3 | 10 | 5
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4 | 2 | 1 | 1 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 14 | 7 | 4 | 10 | 9 | 2
PYREXIA (General disorders) | 17 | 11 | 7 | 6 | 6 | 5
RASH (Skin and subcutaneous tissue disorders) | 24 | 9 | 6 | 16 | 12 | 3
TACHYCARDIA (Cardiac disorders) | 4 | 1 | 0 | 0 | 0 | 3
VOMITING (Gastrointestinal disorders) | 19 | 14 | 13 | 5 | 5 | 4
ASTHENIA (General disorders) | 14 | 20 | 11 | 4 | 7 | 8
CHILLS (General disorders) | 4 | 1 | 6 | 2 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 16 | 18 | 12 | 9 | 8 | 8
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 4 | 0 | 2 | 0 | 0 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 11 | 15 | 15 | 11 | 8 | 6
OEDEMA PERIPHERAL (General disorders) | 8 | 6 | 6 | 0 | 3 | 4
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 1 | 8 | 0 | 4 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 5 | 3 | 4 | 5 | 0
CHEST PAIN (General disorders) | 9 | 8 | 11 | 4 | 12 | 9
DRY SKIN (Skin and subcutaneous tissue disorders) | 4 | 5 | 1 | 1 | 0 | 1
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 4 | 4 | 3 | 4
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 3 | 7 | 7 | 1 | 2 | 6
PAIN (General disorders) | 7 | 8 | 7 | 3 | 6 | 5
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 4 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 10 | 13 | 12 | 5 | 6 | 7
ANXIETY (Psychiatric disorders) | 2 | 2 | 7 | 1 | 1 | 1
DIARRHOEA (Gastrointestinal disorders) | 21 | 20 | 14 | 12 | 14 | 7
DYSGEUSIA (Nervous system disorders) | 7 | 2 | 3 | 0 | 2 | 1
DYSPEPSIA (Gastrointestinal disorders) | 5 | 1 | 4 | 1 | 0 | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 5 | 1 | 6 | 1 | 2 | 1
BONE PAIN (Musculoskeletal and connective tissue disorders) | 5 | 5 | 6 | 4 | 4 | 6
DEPRESSION (Psychiatric disorders) | 4 | 2 | 2 | 0 | 0 | 2
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 1 | 4 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 21 | 11 | 17 | 16 | 12 | 17
FATIGUE (General disorders) | 26 | 24 | 24 | 15 | 15 | 19
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 | 6 | 5 | 1 | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 6 | 4 | 7 | 6 | 4 | 2
NEUROPATHY PERIPHERAL (Nervous system disorders) | 12 | 10 | 19 | 6 | 12 | 5
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4 | 2 | 2 | 1
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 | 0 | 3 | 0 | 3 | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 7 | 14 | 9 | 10 | 15 | 14
ALOPECIA (Skin and subcutaneous tissue disorders) | 27 | 32 | 31 | 24 | 29 | 28
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 | 6 | 9 | 2 | 3 | 3
HYPONATRAEMIA (Metabolism and nutrition disorders) | 3 | 2 | 4 | 1 | 1 | 0
INSOMNIA (Psychiatric disorders) | 8 | 5 | 5 | 2 | 3 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 11 | 9 | 2 | 3 | 5 | 5
PNEUMONIA (Infections and infestations) | 7 | 1 | 1 | 3 | 1 | 0
STOMATITIS (Gastrointestinal disorders) | 1 | 1 | 0 | 4 | 1 | 3
VISION BLURRED (Eye disorders) | 5 | 2 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.